CLINICAL TRIAL: NCT04432441
Title: Effects of Neuromuscular Electrical Stimulation (NMES) Plus Therapeutic Exercise Combination on Scapular Stability in Female Professional Handball Players With Scapular Dyskinesia
Brief Title: Effects of Neuromuscular Electrostimulation on Scapular Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Collaborators: Luis Espejo Antúnez (Unknown); Antoni Morral (Unknown)
Responsible Party: Principal Investigator, Javier Gutiérrez Coronado, Principal Investigator, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19741974
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Adult Female Handball Player
Keywords: "Electric Stimulation Therapy"; "Resistance training"; "Overhead sports"; "Risk factors"; "Scapular anomalies"

STUDY DESIGN:
Intervention Model Description: Two groups. Experimental group realizes a therapeutic physical exercise program for scapulo-humeral stabilitation, and the other group (control group) the same program with electrostimulation. The programme consisted of a two-part sequence of isometric prone push-up, being it an optimal position for periscapular stability exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic physical exercise program for scapulo-humeral stabilitation (Active Comparator): Therapeutic physical exercise program for scapulo-humeral stabilitation
  Interventions: Other: Therapeutic physical exercise program for scapulo-humeral stabilitation
- Therapeutic physical exercise program for scapulo-humeral stabilitation + Electrostimulation (Active Comparator): Therapeutic physical exercise program for scapulo-humeral stabilitation + Electrostimulation
  Interventions: Other: Therapeutic physical exercise program for scapulo-humeral stabilitation + electrostimulation

INTERVENTIONS:
Other: Therapeutic physical exercise program for scapulo-humeral stabilitation — This group realize a therapeutic physical exercise program for scapulo-humeral stabilitation during a month
  Arms: Therapeutic physical exercise program for scapulo-humeral stabilitation
Other: Therapeutic physical exercise program for scapulo-humeral stabilitation + electrostimulation — This group realize a therapeutic physical exercise program for scapulo-humeral stabilitation added electrostimulation during a month
  Arms: Therapeutic physical exercise program for scapulo-humeral stabilitation + Electrostimulation

SUMMARY:
Injuries and shoulder pain are common problems in handball, more often among female athletes. The impact on performance and participation shows the need to work on the risk factors to minimize the damage. It has been found an association between scapular dysfunction and pain in the shoulder. Currently there are many exercise programs, but few with electrotherapy implemented. The aim of the study is to assess the effect of a therapeutic physical exercise program for scapulo-humeral stabilitation with and without electrotherapy on scapular stability, glenohumeral internal rotation and external rotation strength.

ELIGIBILITY:
Inclusion Criteria:

* To have more than 18 YO
* To be female
* To do at least 5 hour of sport training per week in last two years
* To be part of federated club that allows them in their weekly practice to participate in recreational matches or small local championship during weekends.
* To have scapular diskinesis by McClure scale

Exclusion Criteria:

* To have an actual injury
* To have an history of injury in last 12 months
* To take drugs that can affect to control motor.
* To be part or participate in a control motor program or specific prevention program
* To have a recent surgery in last year in upper or back.
* A score below 45 points on the Personal Psychological Apprehension Scale.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Scapular Static Positioning Assessment: Upper distance | Changes from baseline after a month
  cm
Scapular Static Positioning Assessment: Lower distance | Changes from baseline after a month
  cm

SECONDARY OUTCOMES:
RI Range of movement | Changes from baseline after a month
  Degrees
External rotation strenght | Changes from baseline after a month
  kg

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No